CLINICAL TRIAL: NCT02623738
Title: A Phase II/III Randomized, Double-masked, Controlled, Parallel Group, Multicenter Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension -AYAME Study-
Brief Title: A Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension -AYAME Study-
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01171503
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo ophthalmic solution (Placebo Comparator): Eyedrop
  Interventions: Drug: Placebo ophthalmic solution
- DE-117 ophthalmic solution low (Experimental): Eyedrop
  Interventions: Drug: DE-117 ophthalmic solution low
- DE-117 ophthalmic solution high (Experimental): Eyedrop
  Interventions: Drug: DE-117 ophthalmic solution high
- Latanoprost ophthalmic solution 0.005% (Active Comparator): Eyedrop
  Interventions: Drug: Latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: Placebo ophthalmic solution
  Arms: Placebo ophthalmic solution
Drug: DE-117 ophthalmic solution low
  Arms: DE-117 ophthalmic solution low
Drug: DE-117 ophthalmic solution high
  Arms: DE-117 ophthalmic solution high
Drug: Latanoprost ophthalmic solution 0.005%
  Other Names: Latanoprost
  Arms: Latanoprost ophthalmic solution 0.005%

SUMMARY:
The purposes of this study are to determine the optimal concentration of DE-117 ophthalmic solution compared to the placebo ophthalmic solution and to determine if intraocular pressure reduction after 4 weeks of treatment with DE-117 ophthalmic solution is non-inferior to latanoprost ophthalmic solution 0.005%.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma or ocular hypertension

Exclusion Criteria:

* Patients at risk of progression of visual field loss
* Patients with severe visual field defect
* Patients with any diseases that preclude participation in this study for safety reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-12-06 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Osaka, Japan

REFERENCES:
- [Derived] Aihara M, Lu F, Kawata H, Iwata A, Odani-Kawabata N, Shams NK. Omidenepag Isopropyl Versus Latanoprost in Primary Open-Angle Glaucoma and Ocular Hypertension: The Phase 3 AYAME Study. Am J Ophthalmol. 2020 Dec;220:53-63. doi: 10.1016/j.ajo.2020.06.003. Epub 2020 Jun 10. PMID 32533949